CLINICAL TRIAL: NCT01320982
Title: A Randomized Trial Administering Minocycline, Acetylsalicylic Acid or Pramipexole vs Placebo as add-on to Antipsychotics in Patients With Schizophrenia or Schizoaffective Disorder
Brief Title: Minocycline, Acetylsalicylic Acid or Pramipexole vs Placebo in Patients With Schizophrenia or Schizoaffective Disorder
Acronym: MAP-S-01
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Mark Weiser MD (PI), Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SHEBA-8273-10-MW-CTIL
Record Dates: First submitted 2011-02-02; First posted 2011-03-23 (Estimated); Last update posted 2011-03-23 (Estimated); Status verified 2011-03

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Schizophrenia; schizoaffective disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Minocycline; Pramipexole; Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- minocycline (Active Comparator): minocycline
  Interventions: Drug: minocycline
- pramipexole (Active Comparator): pramipexole
  Interventions: Drug: pramipexole
- acetylsalicylic acid (Active Comparator): acetylsalicylic acid
  Interventions: Drug: acetylsalicylic acid
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: minocycline — minocycline 100 mg/bid
  Arms: minocycline
Drug: pramipexole — pramipexole 0.125, 0.25, 0.5 and 0.75 mg/bid
  Arms: pramipexole
Drug: acetylsalicylic acid — acetylsalicylic acid 500mg/ bid
  Arms: acetylsalicylic acid
Drug: placebo — placebo bid
  Arms: Placebo

SUMMARY:
The objective of the study is to evaluate the efficacy of Pramipexole, Minocycline and Aspirin compared to placebo, as add-on to anti-psychotics in the treatment of patients with schizophrenia.

DETAILED DESCRIPTION:
Inflammatory processes have been implicated as a cause of schizophrenia (Fan, Goff et al. 2007), and the COX-2 inhibitor, Celecoxib, has been shown to reduce symptoms of schizophrenia (Muller, Krause et al. 2010). Aspirin, which is also a non-steroidal anti-inflammatory drug(NSAID), irreversibly inhibits Cyclooxygenase-1 (COX-1) and modifies the enzymatic activity of Cyclooxygenase-2 (COX-2), thus inhibiting the formation of prostaglandins and reduces inflammatory reaction. In a study funded by the Stanley Medical Research Institute (SMRI) recently published, Laan at all (Laan, Grobbee et al. 2010) administered add-on 1000mg/d of Aspirin to patients with schizophrenia receiving anti-psychotics, and reported reductions in Positive and negative syndrome scale (PANSS) total and PANSS positive scores without substantial side effects.

Minocycline is a second-generation tetracycline that exerts anti-inflammatory and antimicrobial effects while having a distinct neuroprotective profile. Minocycline effects the glutaminergic system, through inhibition of neuronal nitric oxide synthase (nNOS) and blocking of nitric oxide (NO)- induced neurotoxicity (Du et al, 1998; Jiang et al., 2005), and thus has been suggested as a potential treatment for schizophrenia. One published study (Levkovitz, Mendlovich et al. 2010), and another, unpublished study by Bill Deakin found that add-on treatment of 200mg/d of Minocycline was beneficial for symptoms and cognition in schizophrenia, and a study by Miayoka et al (Miyaoka, Yasukawa et al. 2008) administered open-label 450 mg/day Minocycline, and found improvement on positive symptoms.

Indirect pharmacological evidence suggests a relative excess of dopaminergic activity as being implicated in the pathogenesis of some of the symptoms of schizophrenia, and all effective antipsychotics effect dopamine D2 receptors. Pramipexole is a pre-synaptic dopamine auto-receptor agonist hypothesized to improve in symptoms in schizophrenia patients. In an open label study, Kasper at all (Kasper, Barnas et al. 1997) showed statistically significant improvement in PANSS scores in patients not stabilized on haloperidol. Other data indicate that add-on Pramipexole improves symptoms of depression and cognition, in patients with affective disorders (Goldberg, Frye et al. 1999; Sporn, Ghaemi et al. 2000; Goldberg, Burdick et al. 2004; Zarate, Payne et al. 2004), and Malhotra et al, unpublished data.

All of these studies were relatively small, and were performed by investigators with an interest in the compound. The objective of this study is to replicate them in large trial by investigators with no specific interest in the compounds. This proposed study is a multi-arm study, in which patients will be randomized to one of the three study drugs: Pramipexole, Minocycline and Aspirin, or placebo as part of the same protocol. A design by which several active compounds are all compared to the same placebo arm has been utilized before for schizophrenia (Meltzer, Arvanitis et al. 2004). This design has several advantages: in addition to reduced costs and time it exposes fewer patients to placebo, and enables direct comparison between the compounds and not only to the placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18-65 years of age, inclusive
2. Females who are abstinent or practicing an established method of birth control (oral contraceptive tablets, hormonal implant device, hormone patch, injectable contraceptive, intrauterine device.
3. Willing and able to provide informed consent, after the nature of the study has been fully explained
4. Current DSM-IV-TR diagnosis of schizophrenia or schizoaffective disorder as confirmed by modified Structured Clinical Interview for DSM Disorders (SCID) and having had at least 2 prior schizophrenic episodes, or continually ill for at least 6 months.
5. Symptoms: 4 (moderate) or above on Clinical Global Impression scale (CGI-S)and 4 (moderate)or above score on two of the following four Positive and negative syndrome scale (PANSS) items: delusions, hallucinatory behaviors, conceptual disorganization or suspiciousness/ persecution, and/or a total PANSS negative symptoms score of 18.
6. Must be on any antipsychotic drug, for at least 2 weeks prior to the baseline visit, at doses within the Patient Outcome Research Team (PORT) criteria, whenever possible. Patients receiving higher doses will have their records reviewed to insure that their dose is required and, if possible, will be stabilized on a lower dose prior to study entry.
7. Inpatients or outpatients. Inpatients will be randomized 3 days or more after admission

Exclusion Criteria:

1. Unwilling or unable, in the opinion of the Investigator, to comply with study instructions
2. Pregnant or breast-feeding
3. Unstable medical disease (malignancy, poorly controlled diabetes, active ischemic cardiac disease, or cardiomyopathy, serious pulmonary disease, kidney disease, impaired liver functioning. History of hemorrhagic CVA or peptic ulcer disease.
4. Patients treated with: any of the trial medications i.e. pramipexole/minocycline/ acetylsalicylic acid, NSAIDs, anti-coagulants, sucralfate, cimetidine, amantadine, mexiletine.
5. Likely allergy or sensitivity to raloxifene/pramipexole/minocycline/acetylsalicylic acid.
6. At significant risk of committing suicide, or in the opinion of the Investigator, currently is at imminent risk of suicide or harming others.
7. Patients with a current DSM-IV substance or alcohol abuse. Patients with a history of and/or current recreational use of cannabinoids or alcohol, and/or patients who smoke cigarettes can be included.
8. Concurrent delirium, mental retardation, drug-induced psychosis, or history of clinically significant brain trauma documented by CT or MRI.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-06 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS)total score | Positive and Negative Syndrome Scale (PANSS) total score at week 8
  Change from baseline in Positive and Negative Syndrome Scale (PANSS)total score at 8 weeks
Positive and Negative Syndrome Scale (PANSS)total score | Positive and Negative Syndrome Scale (PANSS) total score at week 16
  Change from baseline in Positive and Negative Syndrome Scale (PANSS)total score at 16 weeks.

SECONDARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS) | Positive and Negative Syndrome Scale (PANSS)positive sub-scale score at week 2
  Change from baseline in Positive and negative syndrome scale(PANSS) positive sub-scale scoreat 2 weeks.
Positive and Negative Syndrome Scale (PANSS) | Positive and Negative Syndrome Scale(PANSS) positive sub-scale score at week 4 .
  Change from baseline in Positive and Negative Syndrome Scale(PANSS) positive sub-scale score at 4 weeks.
Positive and Negative Syndrome Scale (PANSS) | Positive and negative syndrome scale(PANSS) positive sub-scale score at week 8.
  Change from baseline in Positive and negative syndrome scale(PANSS) positive sub-scale score at 8 weeks.
Positive and Negative Syndrome Scale (PANSS) | Positive and negative syndrome scale(PANSS) positive sub-scale score at week 16.
  Change from baseline in Positive and negative syndrome scale(PANSS) positive sub-scale score at 16 weeks.
Positive and Negative Syndrome Scale (PANSS) | Positive and Negative Syndrome Scale (PANSS) negative sub-scale score at week 2
  Change from baseline in Positive and Negative Syndrome Scale (PANSS) negative sub-scale score at 2 weeks
Positive and Negative Syndrome Scale (PANSS) | Positive and Negative Syndrome Scale (PANSS) negative sub-scale score at week 4
  Change from baseline in Positive and Negative Syndrome Scale (PANSS) negative sub-scale score at 4 weeks
Positive and Negative Syndrome Scale (PANSS) | Positive and Negative Syndrome Scale (PANSS) negative sub-scale score at week 8
  Change from baseline in Positive and Negative Syndrome Scale (PANSS) negative sub-scale score at 8 weeks
Positive and Negative Syndrome Scale (PANSS) | Positive and Negative Syndrome Scale (PANSS) negative sub-scale score at week 16
  Change from baseline in Positive and Negative Syndrome Scale (PANSS) negative sub-scale score at 16 weeks
Positive and Negative Syndrome Scale (PANSS) | Positive and Negative Syndrome Scale (PANSS) general psychopathology sub-scale score at 2 weeks
  Change from baseline in Positive and Negative Syndrome Scale (PANSS) general psychopathology sub-scale score at week 2
Positive and Negative Syndrome Scale (PANSS) | Positive and Negative Syndrome Scale (PANSS) general psychopathology sub-scale score at week 4
  Change from baseline in Positive and Negative Syndrome Scale (PANSS) general psychopathology sub-scale score at 4 weeks
Positive and Negative Syndrome Scale (PANSS) | Positive and Negative Syndrome Scale (PANSS) general psychopathology sub-scale score at week 8
  Change from baseline in Positive and Negative Syndrome Scale (PANSS) general psychopathology sub-scale score at 8 weeks
Positive and Negative Syndrome Scale (PANSS) | Positive and Negative Syndrome Scale (PANSS) general psychopathology sub-scale score at week 16
  Change from baseline in Positive and Negative Syndrome Scale (PANSS) general psychopathology sub-scale score at 16 weeks
Clinical Global Impression Scale-Severity (CGI-S) | Clinical Global Impression Scale-Improvement (CGI-S) at week 2
  Change from baseline in Clinical Global Impression Scale-Severity(CGI-S)at 2 weeks
Clinical Global Impression Scale-Severity (CGI-S) | Clinical Global Impression Scale-Severity (CGI-S) at week 5
  Change from baseline in Clinical Global Impression Scale-Severity(CGI-S)at 5 weeks
Clinical Global Impression Scale-Severity(CGI-S) | linical Global Impression Scale-Severity(CGI-S) at week 8
  Change from baseline in Clinical Global Impression Scale-Severity(CGI-S)at 8 weeks
Clinical Global Impression Scale-Severity(CGI-S) | Change from baseline in Clinical Global Impression Scale-Severity(CGI-S) at week 12
  Change from baseline in Clinical Global Impression Scale-Severity(CGI-S)at 12 weeks
Clinical Global Impression Scale-Severity(CGI-S) | Change from baseline in Clinical Global Impression Scale-Severity(CGI-S) at week 16
  Change from baseline in Clinical Global Impression Scale-Severity(CGI-S)at 16 weeks
Clinical Global Impression Scale- Improvement (CGI-I) | Clinical Global Impression Scale- Improvement (CGI-I) at week 2
  Change from baseline in Clinical Global Impression Scale- Improvement (CGI-I)at 2 weeks
Clinical Global Impression Scale- Improvement (CGI-I) | Clinical Global Impression Scale- Improvement (CGI-I) at week 5
  Change from baseline in Clinical Global Impression Scale- Improvement (CGI-I)at 5 weeks
Clinical Global Impression Scale- Improvement (CGI-I) | Clinical Global Impression Scale- Improvement (CGI-I)at week 8
  Change from baseline in Clinical Global Impression Scale- Improvement (CGI-I)at 8 weeks
Clinical Global Impression Scale- Improvement (CGI-I) | Clinical Global Impression Scale- Improvement (CGI-I) at week 12
  Change from baseline in Clinical Global Impression Scale- Improvement (CGI-I)at 12 weeks
Clinical Global Impression Scale- Improvement (CGI-I) | Clinical Global Impression Scale- Improvement (CGI-I)at week 16
  Change from baseline in Clinical Global Impression Scale- Improvement (CGI-I)at 16 weeks
Brief Assessment of Cognition in Schizophrenia (BACS) | rief Assessment of Cognition in Schizophrenia (BACS)at week 8
  Change from baseline in Brief Assessment of Cognition in Schizophrenia (BACS)at 8 weeks.
Brief Assessment of Cognition in Schizophrenia (BACS) | Brief Assessment of Cognition in Schizophrenia (BACS)at week 16
  Change from baseline in Brief Assessment of Cognition in Schizophrenia (BACS)at 16 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Weiser, MD, Principal Investigator — Sheba Medical Center
Locations (7):
- Sheba Medical Center, Ramat Gan, Israel
- Romania (6):
  - Clinica de Psihiatrie, Arad
  - Spitalul de Psihiatrie Botosani, Sectia Psihiatrie, Botoșani
  - Spitalul Clinic de Psihiatrie "Prof. Dr. Alex. Obregia", Bucharest
  - Sp. Jud. "Prof. Dr.O. Fodor", Cluj-Napoca
  - Spitalul Clinic Judetean de Urgenta Cluj, Cluj-Napoca
  - Spitalul Clinic de Psihiatrie Socola, Iasi, Iași

REFERENCES:
- [Derived] Levi L, Zamora D, Nastas I, Gonen I, Radu P, Matei V, Ciobanu AM, Nacu A, Boronin L, Karakrah L, Davidson M, Davis JM, Weiser M. Add-On Pramipexole for the Treatment of Schizophrenia and Schizoaffective Disorder: A Randomized Controlled Trial. J Clin Psychiatry. 2022 Aug 1;83(5):21m14233. doi: 10.4088/JCP.21m14233. PMID 35921506
- [Derived] Weiser M, Zamora D, Levi L, Nastas I, Gonen I, Radu P, Matei V, Nacu A, Boronin L, Davidson M, Davis JM. Adjunctive Aspirin vs Placebo in Patients With Schizophrenia: Results of Two Randomized Controlled Trials. Schizophr Bull. 2021 Jul 8;47(4):1077-1087. doi: 10.1093/schbul/sbaa198. PMID 33479775